CLINICAL TRIAL: NCT07370363
Title: Effects of Moderate-Intensity Continuous Exercise Versus Brisk Interval Exercise on Cardiometabolic Parameters and Sestrin-2 Levels in Hypertensive Obese Women: A Randomized Controlled Trial
Brief Title: Exercise Effects on Cardiometabolic Health and Sestrin-2 in Hypertensive Obese Women
Acronym: SES-EX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Havva Talay Çalış (Other Government)
Responsible Party: Sponsor-Investigator, Havva Talay Çalış, Professor of Physical Medicine and Rehabilitation, Kayseri City Hospital
Organization: Kayseri City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KayseriCHsestrin2
Record Dates: First submitted 2026-01-04; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Hypertension
Keywords: Hypertension; obesity; VO2max; Cardiopulmonary Exercise Testing; Sestrin-2; Aerobic Exercise
MeSH Terms: conditions — Obesity; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Intensity Continuous Exercise (Experimental): Participants perform supervised moderate-intensity continuous aerobic exercise at a prescribed intensity and frequency.
  Interventions: Behavioral: Moderate-Intensity Continuous Exercise
- Brisk Interval Exercise (Experimental): Participants perform supervised interval aerobic exercise consisting of alternating bouts of higher and moderate intensity.
  Interventions: Behavioral: Brisk Interval Exercise

INTERVENTIONS:
Behavioral: Moderate-Intensity Continuous Exercise — Supervised moderate-intensity continuous aerobic exercise performed at a prescribed intensity and frequency for the duration of the intervention period.
  Arms: Moderate-Intensity Continuous Exercise
Behavioral: Brisk Interval Exercise — Supervised interval aerobic exercise consisting of alternating bouts of higher and moderate intensity performed throughout the intervention period.
  Arms: Brisk Interval Exercise

SUMMARY:
Obesity is a chronic and complex disease characterized by excessive fat accumulation that adversely affects health and quality of life. It is commonly accompanied by low-grade chronic systemic inflammation, which contributes to the development of insulin resistance, type 2 diabetes, dyslipidemia, hypertension, and cardiovascular diseases. Hypertension is highly prevalent among individuals with obesity, and excess body weight is a major contributor to elevated blood pressure and related cardiometabolic risk.

Regular aerobic exercise is a cornerstone of non-pharmacological management for both obesity and hypertension and has been shown to reduce chronic inflammation by downregulating pro-inflammatory pathways and upregulating anti-inflammatory mechanisms. Sestrin-2, a stress-responsive protein encoded by the SESN2 gene, has been proposed as an important regulator of metabolic homeostasis and inflammation through activation of the AMPK pathway and inhibition of NF-κB signaling. However, evidence regarding the effects of different exercise modalities on circulating Sestrin-2 levels in hypertensive obese individuals remains limited.

This prospective, randomized controlled trial aims to compare the effects of two different aerobic exercise protocols on serum Sestrin-2 levels, inflammatory status, and cardiometabolic parameters in hypertensive obese women. Cardiopulmonary exercise testing will be used to comprehensively assess cardiorespiratory fitness and physiological responses to exercise. The results of this study are expected to contribute to a better understanding of exercise-induced anti-inflammatory mechanisms and to support the development of safe, effective, and applicable exercise prescriptions for hypertensive obese women.

DETAILED DESCRIPTION:
Obesity is a chronic disease associated with excessive adipose tissue accumulation and a persistent low-grade inflammatory state, which contributes to the development of cardiometabolic disorders such as hypertension, insulin resistance, dyslipidemia, and cardiovascular disease. In women, the coexistence of obesity and hypertension substantially increases morbidity and negatively affects functional capacity and quality of life. Exercise training is a cornerstone of lifestyle-based management; however, the optimal characteristics of aerobic exercise prescription and its effects on emerging molecular biomarkers remain incompletely understood.

Sestrin-2 is a stress-inducible protein encoded by the SESN2 gene and has been implicated in metabolic regulation through activation of the AMP-activated protein kinase pathway and suppression of inflammatory signaling pathways, including nuclear factor kappa B. Experimental and clinical evidence suggests that Sestrin-2 may play a protective role against obesity-related inflammation and metabolic dysfunction. Nevertheless, data regarding the modulation of circulating Sestrin-2 levels in response to different aerobic exercise modalities in hypertensive obese women are limited.

This study is designed as a prospective, randomized controlled trial including hypertensive obese women who meet predefined eligibility criteria. Participants are randomly allocated to one of two supervised aerobic exercise intervention groups: moderate-intensity continuous exercise or brisk interval exercise. Both interventions are conducted for a predefined training period under standardized conditions.

Cardiopulmonary exercise testing is performed to assess cardiorespiratory fitness and physiological responses to exercise, including maximal oxygen consumption. Blood samples are collected to measure serum Sestrin-2 levels and cardiometabolic parameters. Additional assessments include lipid profile, indices of insulin resistance, anthropometric measurements, functional capacity evaluated by the six-minute walk test, and patient-reported questionnaire outcomes.

The primary outcome measures of the study are changes in serum Sestrin-2 levels and maximal oxygen consumption. Secondary outcome measures include changes in cardiometabolic risk factors, functional capacity, and anthropometric parameters. The findings of this study are expected to provide insight into exercise-induced anti-inflammatory mechanisms and to inform evidence-based aerobic exercise prescriptions for hypertensive obese women.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged between 30 and 65 years
* Body mass index between 30.0 and <40.0 kg/m² (Class I and Class II obesity)
* Diagnosis of hypertension according to the 2018 European Society of Hypertension/European Society of Cardiology (ESH/ESC) guidelines
* Sedentary lifestyle, defined as total weekly exercise duration of less than 60 minutes
* Medically eligible for exercise participation, with approval from a Physical Medicine and Rehabilitation specialist and an Internal Medicine specialist
* Willingness to participate in the study and provision of written informed consent

Exclusion Criteria:

* Neuromuscular disorders, uncontrolled psychiatric diseases, or cognitive impairment limiting exercise participation
* Congestive heart failure, unstable angina, or acute cardiac conditions including acute myocardial infarction, acute endocarditis, myocarditis, or pericarditis
* Presence of uncontrolled systemic diseases, including:
* Uncontrolled hypertension
* Uncontrolled diabetes mellitus
* Chronic liver failure
* Chronic kidney disease or patients receiving dialysis
* Chronic obstructive pulmonary disease or asthma
* History or presence of malignancy
* Acute infection at the time of enrollment
* Acute peripheral vascular disease
* Symptomatic severe aortic stenosis
* Acute pulmonary embolism or pulmonary infarction
* Use of systemic corticosteroids or immunosuppressive medications
* Inability to comply with the study protocol or lack of cooperation
* Refusal to participate in the study

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Serum Sestrin-2 Level | Baseline and end of 8-week intervention
  Serum Sestrin-2 levels will be measured using enzyme-linked immunosorbent assay (ELISA).
  Blood samples will be collected 48 hours before the start of the 8-week exercise program and 48 hours after completion of the intervention in order to avoid the acute effects of exercise.
  The primary outcome is the change in Sestrin-2 levels from baseline to post-intervention.
Maximal Oxygen Consumption (VO2max) | Baseline and end of 8-week intervention
  VO2max will be assessed using cardiopulmonary exercise testing (CPET) according to standardized protocols.
  Measurements will be performed before the start of the exercise program and after completion of the 8-week intervention.
  The change in VO2max from baseline to post-intervention will be analyzed.

SECONDARY OUTCOMES:
Lipid Profile | Baseline and end of 8-week intervention
  Fasting blood samples will be collected to assess lipid profile parameters, including total cholesterol, low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and triglyceride levels.
  Standard laboratory methods will be used for biochemical analysis. Changes in lipid profile parameters from baseline to the end of the 8-week exercise intervention will be evaluated.
Insulin Resistance | Baseline and end of 8-week intervention
  Insulin resistance will be assessed using the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR).
  Fasting plasma glucose and fasting insulin levels will be measured using standard laboratory methods, and HOMA-IR will be calculated accordingly.
  The change in HOMA-IR from baseline to the end of the 8-week exercise intervention will be analyzed.
Functional Capacity | Baseline and end of 8-week intervention
  Functional exercise capacity will be assessed using the 6-minute walk test (6MWT) according to established guidelines.
  The total distance walked in six minutes will be recorded at baseline and after completion of the 8-week exercise intervention.
  The change in 6-minute walk distance from baseline to post-intervention will be analyzed.
Blood Pressure | Baseline and end of 8-week intervention
  Resting systolic and diastolic blood pressure will be measured using a validated automated sphygmomanometer according to standardized guidelines.
  Measurements will be performed after at least 5 minutes of seated rest at baseline and after completion of the 8-week exercise intervention.
  The change in systolic and diastolic blood pressure from baseline to post-intervention will be analyzed.
Change in body weight | Baseline and Week 8
  Body weight will be measured in kilograms using a calibrated digital scale at baseline and after completion of the 8-week exercise intervention.
  The change in body weight from baseline to post-intervention will be analyzed.
Change in body mass index (BMI) | Baseline and Week 8
  Body mass index (BMI) will be calculated as weight in kilograms divided by height in meters squared (kg/m²).
  BMI will be assessed at baseline and after completion of the 8-week exercise intervention.
  The change in BMI from baseline to post-intervention will be analyzed.
Change in waist circumference | Baseline and Week 8
  Waist circumference will be measured in centimeters using a non-elastic measuring tape according to standardized procedures.
  Measurements will be performed at baseline and after completion of the 8-week exercise intervention.
  The change in waist circumference from baseline to post-intervention will be analyzed.
Change in International Physical Activity Questionnaire (IPAQ) score | Baseline and Week 8
  Physical activity levels will be assessed using the International Physical Activity Questionnaire (IPAQ).
  The IPAQ provides physical activity estimates expressed as metabolic equivalent task minutes per week (MET-min/week), with higher values indicating higher physical activity levels.
  The questionnaire will be administered at baseline and after completion of the 8-week exercise intervention.
  The change in IPAQ score from baseline to post-intervention will be analyzed.
Change in Hospital Anxiety and Depression Scale (HADS) scores | Baseline and Week 8
  Anxiety and depressive symptoms will be assessed using the Hospital Anxiety and Depression Scale (HADS).
  The HADS consists of 14 items and includes two subscales: anxiety (HADS-A) and depression (HADS-D), each scored from 0 to 21.
  Higher scores indicate greater levels of anxiety or depressive symptoms. The questionnaire will be administered at baseline and after completion of the 8-week exercise intervention.
  Changes in HADS-A and HADS-D scores from baseline to post-intervention will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JH, Budanov AV, Karin M. Sestrins orchestrate cellular metabolism to attenuate aging. Cell Metabolism. 2013;18(6):792-801.
- [Background] Williams B, Mancia G, Spiering W, et al. 2018 ESC/ESH Guidelines for the management of arterial hypertension. European Heart Journal. 2018;39(33):3021-3104.